CLINICAL TRIAL: NCT04723537
Title: Phase 2/3 Study of Upamostat, a Serine Protease Inhibitor, or Placebo for Treatment of COVID-19 Disease
Brief Title: Upamostat, a Serine Protease Inhibitor, or Placebo for Treatment of COVID-19 Disease
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Part A complete; corporate decision made to cancel Part B.
Sponsor: RedHill Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RHB-107-01
Record Dates: First submitted 2021-01-18; First posted 2021-01-25 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: Upamostat 200 mg (Experimental): Each day participants will receive a single 200 mg dose of upamostat along with a single matching placebo, for a total of 14 days.
  Interventions: Drug: Part A: Upamostat 200 mg
- Part A: Upamostat 400 mg (Experimental): Each day participants will receive two 200 mg doses of upamostat, for a total of 14 days.
  Interventions: Drug: Part A: Upamostat 400 mg
- Part A: Placebo (Placebo Comparator): Each day participants will receive two matching placebos, for a total of 14 days.
  Interventions: Drug: Part A and B: Placebo
- Part B: Upamostat (Experimental): Based on dose selected from Part A, each day participants will receive EITHER a single 200 mg dose of upamostat OR two 200 mg doses of upamostat, for a total of 14 days.
  Interventions: Drug: Part B: Upamostat 200 or 400 mg
- Part B: Placebo (Placebo Comparator): Based on dose selected from Part A, each day participants will receive EITHER a single matching placebo OR two matching placebos, for a total of 14 days.
  Interventions: Drug: Part A and B: Placebo

INTERVENTIONS:
Drug: Part A: Upamostat 200 mg — 1 capsule comprising 200 mg of upamostat and 1 capsule comprising matching placebo.
  Arms: Part A: Upamostat 200 mg
Drug: Part A: Upamostat 400 mg — 2 capsules, each capsule comprising 200 mg of upamostat
  Arms: Part A: Upamostat 400 mg
Drug: Part A and B: Placebo — 1 or 2 capsules, each capsule a matching placebo
  Arms: Part A: Placebo; Part B: Placebo
Drug: Part B: Upamostat 200 or 400 mg — Based on dose selection from Part A, "Part B Upamostat" will be EITHER a single 200 mg dose of upamostat OR two 200 mg doses of upamostat, for a total of 14 days.
  Arms: Part B: Upamostat

SUMMARY:
A 2-part, multicenter, Phase 2/3, randomized, double-blind, placebo-controlled, parallel group study to evaluate the safety and efficacy of upamostat in adult patients with COVID-19 disease who do not require inpatient care.

DETAILED DESCRIPTION:
Patients will be seen in a medical facility (ER or COVID-19 clinic) for initial evaluation. Consenting, diagnostically-confirmed COVID-19 patients not in need of hospitalization per investigator assessment and who meet all other inclusion and exclusion criteria will be randomized to treatment and provided with medication and home monitoring devices, and instructed in drug administration and use of the devices. They will take medication daily for two weeks, complete a smartphone-based questionnaire, provide additional monitoring information via devices provided periodically over an 8-week period. Patients will be seen at home by a study nurse or return to the clinic after 2, 4 and 8 weeks on study ("follow up" visits); additional televisits will also be conducted. At the follow up visits nasal swab specimens for COVID-19 PCR and blood specimens for safety labs and disease markers will be collected.

In part A of the study, patients will be randomized 1:1:1 to one of two doses of upamostat or placebo. Based on safety results of part A, a dose for part B will be selected, and patients will be randomized 3:2 to active vs placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic, diagnostically confirmed COVID-19, per RT-PCR or antigen assay of respiratory tract sample.
2. Patient must have either become symptomatic or found positive by RT-PCR or antigen assay within 5 days, whichever is greater, of randomization.
3. Patients must fill out a baseline questionnaire which is reviewed by study personnel to determine eligibility.
4. Males and females ≥age 18 years.
5. Oxygen saturation by pulse oximeter ≥92% on room air
6. Negative urine or serum pregnancy test (if woman of childbearing potential).
7. Females of childbearing potential and males with female partners of childbearing potential must agree to use acceptable contraceptive methods during the study and for at least two months after the last dose of study medication.
8. Ability to complete the daily diary independently.
9. The patient must give informed consent

Exclusion Criteria:

1. Patient is in need of acute hospitalization per clinician assessment.
2. Pregnant or nursing women.
3. Unwillingness or inability to comply with procedures required in this protocol.
4. Patient requires supplemental oxygen.
5. Patient is currently receiving, has received within the past 7 days or is expected to receive during the course of the study remdesivir, or other specific antiviral or anticytokine therapy for COVID-19, other than therapeutic monoclonal antibodies allowed or approved in the region in which the patient lives, or systemic corticosteroid equivalent to ≥20 mg daily prednisone/3 mg dexamethasone daily.
6. Patient is currently receiving or has received within 30 days prior to screening any other investigational agent for any indication, including approved agents given for investigational indications (e.g., anti-cytokine treatments).
7. Patient is currently taking or is expected to start taking warfarin, apixaban (Eliquis), or rivaroxaban (Xarelto). Patients may be taking or start on study dabigatran (Pradaxa), standard or low molecular weight heparin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry Plasse, MD, Study Director — RedHill Biopharma Limited
Locations (17):
- United States (11):
  - Beautiful Minds Clinical Research, Cutler Bay, Florida
  - Research in Miami Inc., Hialeah, Florida
  - Angels Clinical Research Institute, Miami, Florida
  - South Florida Research Phase I-IV, Inc., Miami Springs, Florida
  - Great Lakes Research Group, Bay City, Michigan
  - Henry Ford Hospital, emergency department, Detroit, Michigan
  - Prime Global Research, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - On-Site Clinical Solutions, Charlotte, North Carolina
  - University Hospitals Cleveland, Cleveland, Ohio
  - Southwest Family Medicine Research, Dallas, Texas
- South Africa (6):
  - Langeberg Medical Centre - Clinical Trials, Kraaifontein, Cape Town
  - Roodepoort Medicross Clinical Trial Research Centre, Roodepoort, Gauteng
  - FCRN Clinical Trial Centre, Vereeniging, Gauteng
  - PJ Sebastian, KwaZulu, KwaZulu-Natal
  - Global Clinical Trials PTY (LTD), Arcadia, Pretoria
  - WorthWhile Clinical Trials, Benoni

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Plasse TF, Delgado B, Potts J, Abramson D, Fehrmann C, Fathi R, McComsey GA. A randomized, placebo-controlled pilot study of upamostat, a host-directed serine protease inhibitor, for outpatient treatment of COVID-19. Int J Infect Dis. 2023 Mar;128:148-156. doi: 10.1016/j.ijid.2022.12.003. Epub 2022 Dec 19. PMID 36549549
- [Result] Plasse TF, Fathi R, Fehrmann C, McComsey GA. Upamostat: a serine protease inhibitor for antiviral, gastrointestinal, and anticancer indications. Expert Opin Investig Drugs. 2023 Jul-Dec;32(12):1095-1103. doi: 10.1080/13543784.2023.2284385. Epub 2023 Dec 28. PMID 37970658

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part A: Upamostat 200 mg | Part A: Upamostat 400 mg | Part A: Placebo
Started | 20 | 21 | 20
Completed | 16 | 20 | 18
Not Completed | 4 | 1 | 2
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Medical monitor decision, sponsor decision and other | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Upamostat 200 mg | Part A: Upamostat 400 mg | Part A: Placebo | Total
Number analyzed (Participants) | 20 | 21 | 20 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 18 | 55
  >=65 years | 2 | 2 | 2 | 6
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40.5 [26.0 to 55.0] | 50.0 [41.0 to 60.0] | 46.0 [33.0 to 53.5] | 47.0 [32.0 to 55.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 11 | 34
  Male | 6 | 12 | 9 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 2 | 6
  White | 18 | 17 | 16 | 51
  More than one race | 1 | 0 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 10 | 10 | 7 | 27
  Non-Hispanic/Non-Latino | 10 | 11 | 13 | 34
Region of Enrollment [Number; unit: participants]
  United States | 19 | 21 | 20 | 61
  South Africa | 1 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A - Determination of the Safety and Tolerability of Two Dose Levels and Selection of an Upamostat Dose for Part B
Description: This is a qualitative measure that takes into account safety and tolerability based on the relative incidence and severity (CTCAE v 5.0 criteria) of adverse events, both clinical and laboratory (SOC=investigations) in each active treatment group as compared to placebo. In addition, toxicities (i.e., adverse events considered at lease possible related to study medication) resulting in dose reductions or discontinuation of therapy will be tabulated and compared among treatment groups.
Time Frame: 57 days
Population: All patients entered
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Upamostat 200 mg | Part A: Upamostat 400 mg | Part A: Placebo
Number analyzed (Participants) | 20 | 21 | 20
Participants
  Safe and well tolerated | 20 | 21 | 20
  Dose reductions or discontinuation of therapy | 0 | 0 | 0

2. Secondary Outcome: Hospitalization or Death From Any Cause by End of Study
Time Frame: 57 days
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Upamostat 200 mg | Part A: Upamostat 400 mg | Part A: Placebo
Number analyzed (Participants) | 20 | 21 | 20
Participants | 0 | 1 | 3

3. Secondary Outcome: Hospitalization or Death For COVID With Presence of Concerning Conditions
Time Frame: 57 days
Population: Patient with concerning conditions per NIAID guideline
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Upamostat 200 mg | Part A: Upamostat 400 mg | Part A: Placebo
Number analyzed (Participants) | 8 | 15 | 13
Participants | 0 | 0 | 2

4. Secondary Outcome: Time to Sustained Recovery From Symptomatic Illness for Part A (Protocol Definition)
Description: Sustained recovery was defined as recovery maintained for at least 14 or 28 days (two analyses), or through end of study, whichever comes first. A patient was considered to have recovered once he or she met the following criteria:
  1. is afebrile (<38.0°C core temperature/37.5°C oral temperature) for at least 48 hours without use of antipyretics;
  2. all symptoms have resolved or returned to pre-illness levels (e.g., if patient had respiratory compromise prior to the onset of COVID), except for:
     1. fatigue, anosmia, ageusia or dysgeusia, which may be persistent at level similar to that during the acute illness, i.e., the same level per symptom questionnaire;
     2. chest pain, cough or dyspnea which if persistent must be at least one grade lower than at the start of treatment and no worse than grade 1 (mild).
Time Frame: 57 days
Population: ITT
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Part A: Upamostat 200 mg | Part A: Upamostat 400 mg | Part A: Placebo
Number analyzed (Participants) | 20 | 21 | 20
days | 19.0 [13.0 to 57.0] | 27.0 [14.0 to 43.0] | 19 [12.5 to 38.0]

5. Secondary Outcome: Time to Sustained Recovery From Symptomatic Illness - Part A (SAP Definition)
Description: First day at which there are no symptoms, and no occurrence of any symptoms for at least 14 days or until end of study, whichever came first. Mild symptoms which were noted as preexisting conditions were excluded from this calculation. For example, if a patient noted preexisting shortness of breath, mild shortness of breath was excluded from the calculation of no symptoms.
Time Frame: 57 days
Population: ITT
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Part A: Upamostat 200 mg | Part A: Upamostat 400 mg | Part A: Placebo
Number analyzed (Participants) | 20 | 21 | 20
days | 29.5 [18.5 to 57.0] | 38.0 [16.0 to 57.0] | 38.0 [15.5 to 57.0]

6. Secondary Outcome: Development of New Disease-related Symptoms and/or Pneumonia on Study
Time Frame: 57 days
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Upamostat 200 mg | Part A: Upamostat 400 mg | Part A: Placebo
Number analyzed (Participants) | 20 | 21 | 20
Participants | 17 | 12 | 16

7. Secondary Outcome: Proportion of Patients Who Are PCR-negative at Day 8 From the Start of Treatment
Time Frame: 8 days
Population: Patients with PCR results
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Upamostat 200 mg | Part A: Upamostat 400 mg | Part A: Placebo
Number analyzed (Participants) | 19 | 19 | 17
Participants | 9 | 10 | 7

8. Secondary Outcome: Proportion of Patients Who Are PCR-negative at Day 57 From the Start of Treatment
Time Frame: 57 days
Population: Patients with PCR results
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Upamostat 200 mg | Part A: Upamostat 400 mg | Part A: Placebo
Number analyzed (Participants) | 16 | 13 | 18
Participants | 16 | 12 | 17

9. Secondary Outcome: Changes in D-dimer Levels, From Baseline to Day 57
Time Frame: 57 days
Population: Patient with D dimer results at end of study
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Part A: Upamostat 200 mg | Part A: Upamostat 400 mg | Part A: Placebo
Number analyzed (Participants) | 14 | 14 | 18
ug/ml | -0.21 (0.27) | -0.64 (0.81) | 0.01 (0.41)

10. Post Hoc Outcome: Time to Sustained Recovery From Severe Symptoms - Part A
Time Frame: 57 days
Population: Patients with severe symptoms at baseline
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Part A: Upamostat 200 mg | Part A: Upamostat 400 mg | Part A: Placebo
Number analyzed (Participants) | 8 | 11 | 10
days | 4.0 [2.0 to 6.0] | 3.0 [2.0 to 6.0] | 8.0 [4.0 to 26.0]

ADVERSE EVENTS:
Time Frame: 57 days
Description: AEs assessed first dose through day 57. All new abnormal lab findings and those abnormal at baseline which change by at least one toxicity grade as defined in [NCI CTCAE] v5.0 were considered AEs.
  Laboratory values outside the normal range will not be considered AEs if they are generally not considered as indicating an abnormality in CTCAE.
  Exacerbation of COVID-19-related signs and symptoms were considered lack of efficacy and not adverse events. Hospitalization for COVID was not an SAE.
Arm/Group | Part A: Upamostat 200 mg | Part A: Upamostat 400 mg | Part A: Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/21 | 0/20
Other Adverse Events (participants affected / at risk) | 19/20 | 20/21 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Upamostat 200 mg (N=20) | Part A: Upamostat 400 mg (N=21) | Part A: Placebo (N=20)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Acute alcohol intoxication in a patient with a history of alcohol abuse
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Upamostat 200 mg (N=20) | Part A: Upamostat 400 mg (N=21) | Part A: Placebo (N=20)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal Refulx Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Application Site Erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Application Site Irritation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Genital Candisiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 7 (7) | 10 (10) | 5 (5)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Albumin Decreased (Investigations) | 1 (1) | 2 (2) | 1 (1)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood Calcium Decreased (Investigations) | 2 (2) | 2 (2) | 1 (1)
Blood Calcium Increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood Carbon Dioxide Decreased (Investigations) | 5 (5) | 0 (0) | 2 (2)
Blood Chloride Decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood Chloride Increased (Investigations) | 7 (7) | 4 (4) | 3 (3)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Glucose Decreased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Blood Glucose Increased (Investigations) | 2 (2) | 2 (2) | 2 (2)
Blood Lactate Dehydrogenase Increased (Investigations) | 2 (2) | 2 (2) | 3 (3)
Blood Potassium Decreased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Blood Potassium Increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Blood Sodium Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Sodium Increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood Urea Nitrogen Increased (Investigations) | 2 (2) | 2 (2) | 3 (3)
C-Reactive Protein Increased (Investigations) | 5 (5) | 3 (3) | 3 (3)
Fibrin D Dimer Increased (Investigations) | 7 (7) | 6 (6) | 6 (6)
Haemoglobin Decreased (Investigations) | 4 (4) | 5 (5) | 2 (2)
Haemoglobin Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
International Normalized Ratio Increased (Investigations) | 10 (10) | 10 (10) | 4 (4)
Lymphocyte Count Decrease (Investigations) | 1 (1) | 0 (0) | 1 (1)
Monocyte Count Increased (Investigations) | 0 (0) | 1 (1) | 3 (3)
Neutrophil Count Decreased (Investigations) | 2 (2) | 2 (2) | 1 (1)
Neutrophil Count Increased (Investigations) | 1 (1) | 3 (3) | 2 (2)
Platelet Count Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet Count Increased (Investigations) | 2 (2) | 1 (1) | 5 (5)
Protein Total Decreased (Investigations) | 7 (7) | 3 (3) | 4 (4)
Protein Total Increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Serum Ferritin Decreased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Serum Ferritin Increased (Investigations) | 1 (1) | 0 (0) | 3 (3)
Transaminases Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Troponin Increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 1 (1) | 4 (4) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash Vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are disclosure agreements between the Sponsor and each of the participating clinical sites and PI that slightly differ.

DOCUMENTS (2):
  • Study Protocol (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT04723537/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT04723537/SAP_001.pdf